CLINICAL TRIAL: NCT06638710
Title: Efficacy and Safety of Oral Midazolam for the Delivery of Care in Elderly Patient With Moderate to Severe Neurocognitive Disorders and Refusing Care
Brief Title: Efficacy and Safety of Oral Midazolam Used for the Delivery of Care in Elderly Patient With Neurocognitive Disorders and Refusing Care.
Acronym: MIRAGE
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Grenoble (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 38RC21.0436
Record Dates: First submitted 2024-09-10; First posted 2024-10-15 (Actual); Last update posted 2025-12-15 (Actual); Status verified 2025-12

CONDITIONS: Neurocognitive Disorders
Keywords: elderly; midazolam; care
MeSH Terms: conditions — Neurocognitive Disorders

STUDY DESIGN:
Intervention Model Description: This is a "n of one design" study
  * Patients presenting opposition to at least two nursing care will be selected for the study.
  * Patients included in the study will be assigned a kit of 20 unit doses containing an oral gel of midazolam or placebo, according to a predefined sequence. Maximum 20 nursing care will be included in the study.
  * For each new opposition to treatment ≥ 3 on the Pittsburgh scale, the nurse will administer the next syringe from the kit in a double-blind manner, following the predefined order. Thirty to forty minutes after administration, the nurse will reassess the level of opposition and then attempt the same care again.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Blinding will be carried out upstream by the pharmacy that will prepare the treatment kits.
  For each nursing treatment, the syringe will contain either midazolam or placebo according to randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo (Placebo Comparator): The nurse administers an oral dose of placebo to the patient
  Interventions: Drug: oral administration of midazolam or placebo
- oral midazolam (Experimental): The nurse administers an oral dose of midazolam to the patient
  Interventions: Drug: oral administration of midazolam or placebo

INTERVENTIONS:
Drug: oral administration of midazolam or placebo — If the patient is opposed to a treatment (resistance to care ≥3 on the Pittsburgh scale), the nurse administers an oral dose of midazolam or placebo to the patient according to the random allocation.

SUMMARY:
The purpose of this study is to assess the effectiveness of oral midazolam on the delivery of care in elderly patients with moderat to severe neurocognitive disorders and opposing care.

DETAILED DESCRIPTION:
Neurodegenerative disorders may lead to behavioral disturbances that can result in oppositional reactions, making the performance of certain medical treatments complex.

Midazolam is used to reduce anxiety and agitation in elderly patients with moderate to severe neurocognitive disorders. It has the advantages of rapid action, short half-life, and good tolerability. A recent study shows that its use by subcutaneous (SC) injection 'as needed,' off-label, is becoming increasingly common in elderly patients, particularly to facilitate care. However, SC injection may be poorly tolerated by patients, difficult to administer, and may cause a feeling of mistreatment.

The aim of this clinical trial is to evaluate the efficacy and safety of an oral form of midazolam adapted for the elderly on the performance of care.

ELIGIBILITY:
Inclusion Criteria:

* Patient hospitalized (for a minimum estimated duration of 21 days) in a geriatric department in Medical Care and Rehabilitation, Cognitive-Behavioral Unit, or housed in a Reinforced Housing Unit, in a Long-Term Care Unit, or in a Psycho-Geriatric Unit.
* Moderate to severe cognitive impairment, defined by a MMSE (Mini Mental State Examination) score <15. If not feasible at inclusion, MMSE score <15 less than 1 year old.
* Patient opposed to care, presenting at least two episodes of opposition to care (meals excluded) for which other non-medication alternatives have failed. These refusals of care are defined by a "resistance to care" score ≥3 on the Pittsburgh scale, over the last week. In practice, the resistance to care of patients is noted in the medical record following a weekly multidisciplinary decision.

The targeted cares:

Essential nursing care (indispensable, mandatory, and prescribed) Bathing and changing made essential by obvious lack of hygiene after evaluation Bedtime installation (e.g., with the SECURIDRAP® device) technical care: blood tests, wound care, dressing changes, insertion of urinary or nasogastric tubes; administration of medication by parenteral route

* Person affiliated with social security or beneficiary of such a scheme
* Informed, written, and signed consent by the patient or their legal representative (for adults under legal protection and unable to express their consent)

Exclusion Criteria:

* Patient who has received midazolam treatment in the week before inclusion
* Patient with contraindications to midazolam:

severe Myasthenia Severe respiratory failure requiring continuous oxygen therapy Severe liver failure: PT <50% Severe sleep apnea syndrome not treated with a device Severe renal failure: Cockcroft <20mL/min Severe heart failure in a state of decompensation History of alcoholism or drug addiction

* Known hypersensitivity to the active substance, benzodiazepines, or any of the excipients
* Patient being treated concurrently with:

CYP3A4 enzyme inhibitors CYP3A4 enzyme inducers

* Weight <50 kg and >100 kg
* Gastrointestinal pathology that may limit or prevent the absorption of midazolam
* Identification of anxiety, defined by item E of the NPI (neuropsychiatric inventory) by an evaluation >2 in frequency and severity according to HAS recommendations.
* Identification of pain, defined by the Algoplus scale by an evaluation ≥2
* Identification of ideational disorders, defined by item E of the Cornell scale: E>0
* Subject in the exclusion period of another clinical trial
* Subject deprived of liberty by an administrative or judicial decision.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-08 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-11-01 (Estimated)

PRIMARY OUTCOMES:
Evolution of resistance to care following oral administration of midazolam | For each care: change of the care dimension of the Pittsburgh scale from the time of intention of care and 30 to 45 minutes after the study treatment intake.
  The efficacy will be evaluated by a decrease of at least two points in the resistance to care dimension of the Pittsburgh scale. the care dimension scale has 4 points, 4 is the worst score, 0 is the better.

SECONDARY OUTCOMES:
effectiveness of oral midazolam in terms of acceptance of care | For each care : This scale is measured immédiately after the end of the care.
  The acceptance of care is evaluated using the care acceptance scale by Rignell et al. (2007). This scale rangin from 1 to 4. the wrongest score is.
Evolution of agitation and refusal to care following oral administration of midazolam | For each care: change from the time of intention of care and 30 to 45 minutes after the study treatment intake.
  Agitation and refusal of care will be evaluated using the global score of the Pittsburgh Agitation Scale. The scale ranging from 0 to 16. the wrongest score is 16
Number and description of Treatment-Related Adverse Events. | From enrollment to the end of treatment at 4 months
  Measurement of saturation, respiratory rate, and heart rate, and collection of serious and non-serious adverse events occurring after the administration of midazolam gel.
Satisfaction of the caregiving staff. | For each care: immediatly after the care.
  Satisfaction questionnaire on the caregivers; sense of well-being towards patients.

CONTACTS AND LOCATIONS:
Locations (1):
- Geriatric department of Grenoble Alpes university hospital, Grenoble, Isere, France

IPD SHARING:
Plan to Share IPD: No